CLINICAL TRIAL: NCT06213766
Title: Joint Analysis of Spatial and Ocular Trajectories for the Early Diagnosis of Alzheimer's Disease.
Brief Title: Spatial and Ocular Trajectories for the Early Diagnosis of Alzheimer's Disease.
Acronym: ACTSOMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL23_1166
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Alzheimer Disease; Aging
Keywords: Alzheimer Disease; spatial navigation; eye-tracking; biomarkers; early diagnosis; personalized medicine; machine learning
MeSH Terms: conditions — Alzheimer Disease; Spatial Navigation; Disease | interventions — Surveys and Questionnaires; Eye-Tracking Technology; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitively healthy subjects (Active Comparator): Participants aged between 20 and 85 years old with no cognitive impairment (Montreal Cognitive Assessment ≥ 26/30 and MacNair Cognitive Difficulties Self-Rating Scale ≥15), affiliated or entitled to a social health insurance, having been informed and having given written consent to the study.
  As part of the study, cognitively healthy subjects will :
  * Undergo a cognitive assessment;
  * Answer several questionnaires on their demographic data, lifestyle habits, quality of sleep, cognitive reserve, concomitant treatment and comorbidities;
  * Complete a cognitive spatial navigation task with eye-tracking;
  * Have a blood sampling for plasma biomarker and genetic risk factor for Alzheimer's disease.
  Interventions: Diagnostic Test: Cognitive assessment; Other: Questionnaires; Device: Spatial navigation task with eye-tracking.; Biological: Blood sampling
- Patients suffering from Alzheimer's disease (Experimental): Patients aged between 50 and 85 years old, undergoing memory clinic consultation for prodromal or mild Alzheimer's disease with mild or moderate cognitive decline (Mini-Mental State Examination ≥20/30) affiliated or entitled to a social health insurance, having been informed and having given written consent to the study.
  As part of the study, patients suffering from Alzheimer's disease will :
  * Undergo a cognitive assessment;
  * Answer several questionnaires on their demographic data, lifestyle habits, quality of sleep, cognitive reserve, concomitant treatment and comorbidities;
  * Complete a cognitive spatial navigation task with eye-tracking;
  * Have a blood sampling for plasma biomarker and genetic risk factor for Alzheimer's disease.
  Interventions: Diagnostic Test: Cognitive assessment; Other: Questionnaires; Device: Spatial navigation task with eye-tracking.; Biological: Blood sampling

INTERVENTIONS:
Diagnostic Test: Cognitive assessment — Group 1: Cognitively healthy subject:
  After signing the consent form, during the only visit of the study, the investigator will administer to cognitively healthy subjects two cognitive screening tests to ensure that they meet the criteria for group 1. If performance on the cognitive scales prove to be borderline or below current standards (Montreal Cognitive Assessment ≥ 26/30 and MacNair Cognitive Difficulties Self-Rating Scale ≥15) for at least one of the 2 tests, the participant will prematurely end the study and may be offered an in-depth cognitive assessment as part of routine care.
  Group 2: Patients suffering from Alzheimer's disease:
  After signing the consent form, during the only visit of the study, the investigator will administer to patients the Montreal Cognitive Assessment to assess cognitive status.
Other: Questionnaires — For every participants (group 1 and 2):
  During the only visit of the study and after the intervention 1, the participants will answer questionnaires about:
  * Demographic data such as age, gender, weight, height, education level;
  * Lifestyle habits such as usual mode of transport, sense of direction, use of GPS device, and video game practice;
  * Quality of sleep over the previous month and the previous night;
  * Cognitive reserve questionnaire from Rami et al., 2011;
  * Concomitant treatment and comorbidities.
Device: Spatial navigation task with eye-tracking. — For every participants (group 1 and 2):
  During the only visit of the study and after interventions 1 and 2, the participants will complete the spatial navigation task with eye-tracking.
  The participants will play the Sea Hero Quest video game and take on the role of the captain of a small boat that has to find its way through an aquatic environment. At the start of each level, the player is shown a map of the environment, with the boat's initial position and the buoys it must reach as quickly as possible in a set order. Once the map has been memorised, it disappears and the navigation begins.
  Participants will play 6 levels of Sea Hero Quest (two training levels and four different navigation levels). This intervention will be proposed by a trained team member and participants will play on a digital tablet connected to an eye-tracker. The total duration of the task is 30 min (training phase + assessment sequences).
Biological: Blood sampling — For every participants (group 1 and 2):
  During the only visit of the study and after interventions 1, 2 and 3, a state-qualified nurse will take venous samples from 3 tubes of 4ml each.
  These blood samples will be frozen and stored until the end of the study when they will be analysed:
  * Sample 1: plasmatic Quanterix p-tau217 assay;
  * Sample 2: apolipoprotein E genotyping;
  * Sample 3: measurement of plasmatic creatinine levels. Neither the cognitively healthy subjects, nor the patients, nor the clinicians in charge of the patients included will be informed of the results of these biological assays (absence of clinical interest established at the present time of the APOE genotype and the p-tau217 protein level, absence of modification of the care pathway, in adequacy to the bioethics law of August 02, 2021. Creatinine level is used in this study as an adjustment variable to interpret the p-tau217 protein level and will not be used for clinical interpretation.

SUMMARY:
Spatial navigation is a high-level cognitive function that enables humans to orientate themselves and move around in space by constructing a mental representation of the environment. It is particularly interesting because it involves numerous neural networks, linked to proprioception and vision, for example.

Despite the versatility of this cognitive function, spatial navigation is little studied clinically, although changes in spatial planning and navigation strategies have been associated with many brain disorders, including Alzheimer's disease (Coughlan et al., 2018). This may be explained in view of the neuropsychological tests currently in use, which do not effectively assess spatial navigation disorders. In addition, many non-pathological parameters - in particular socio-demographic and lifestyle - (Wolbers & Hegarty, 2010; Coutrot et al., 2018) affect spatial navigation performance. Separating the pathological component from these non-pathological factors in spatial navigation can be challenging.

In this context, Sea Hero Quest (SHQ) has been developed (Coutrot et al., 2018; Spiers et al., 2021) as an international-scale cognitive spatial navigation task that holds great promise for assessing spatial navigation performance during normal and pathological ageing. SHQ is a video game that implements classic tasks from the spatial cognition literature, and has enabled the trajectories of 4 million players with varied socio-demographic profiles to be collected.

In addition to the direct measurement of spatial displacements, eye movements, measured by eye-tracking, provide additional information on the cognitive processes associated with visual attention. The analysis of eye movements can provide valuable information about the strategies employed by humans during spatial navigation (Zhu et al., eLife 2023).

While it is well known that normal ageing and pathological ageing (e.g. in the context of Alzheimer's disease) affect performance in simple spatial navigation or visual attention tasks, the neurocognitive mechanisms involved in this deterioration remain poorly understood. The investigators hypothesise that the joint analysis of ocular and spatial traces will provide a more detailed understanding of the cognitive strategies deployed during a spatial navigation task, and therefore of these underlying mechanisms.

The investigators therefore propose to jointly study the association between two complementary cognitive functions: spatial navigation and visual attention, and their relationship with normal and pathological ageing (confirmed Alzheimer's disease, plasma biomarkers and genetic risk factors for Alzheimer's disease). The joint analysis of these different signals has never been carried out as part of research into normal ageing and Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

Cognitively healthy subjects:

* Participants aged between 20 and 85 years old;
* Participant affiliated or entitled to a social security scheme;
* Participants who have been informed and have given written consent.

Patients with Alzheimer's disease:

* Participant aged between 50 to 85 years old;
* Participant undergoing memory clinic consultations for a diagnosed Alzheimer's disease, at the stage of minor neurocognitive impairment or major neurocognitive impairment, according to the NIA-AA 2011 criteria (McKahn et al., 2011, Albert et al., 2011);
* Mild to moderate cognitive impairment, Mini-Mental State Examination (MMSE ≥ 20/30, in the 6 months prior to inclusion);
* Participant affiliated or entitled to a social security scheme;
* Participants who have been informed and have given written consent.

Exclusion Criteria:

For all participants:

* Severe, progressive or unstable pathology whose nature may interfere with the assessment variables (epilepsy, acute psychiatric or psychotic disorders, visual hallucinations, acute infection);
* Consumption of toxic substances that may affect cognitive performance;
* Deafness or blindness that could compromise the participant's assessment or participation in tasks and scales;
* Participants under guardianship or legal protection;
* Pregnant women, women in labour or breastfeeding mothers;
* Persons under psychiatric care.

Cognitively healthy subjects:

- Participants diagnosed with a cognitive disorder.

Specifically for patients with Alzheimer's disease:

* Participants with a diagnosis other than Alzheimer's disease that promotes neurocognitive impairment (with the exception of cerebral microvascular involvement, i.e. mild to moderate microangiopathy);
* Severe cerebral microangiopathy (extensive and severe white matter hypersignals, Fazekas score = 3);
* Severe psycho-behavioral manifestations preventing performance of the task, at the investigator's discretion;
* Current participation in an Alzheimer's disease drug research protocol, in particular testing 'disease-modifying' treatments that may interact with the pathophysiology of the disease (after randomisation).

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of spatial navigation strategies used by participants according to age. | Day 1 Just After inclusion
  Spatial navigation strategies will be described thanks to machine learning identifying spatial navigation patterns taking into consideration:
  * Spatial performances: length of trajectories sampled at 2Hz (1 x-y coordinate every 500 ms) - the shorter the trajectory, the better the performance;
  * Eye movements: gaze sampling recorded and sampled at 60Hz to identify visual clues used by participants to solve the spatial task).
  These patterns will be described according to participant's age.

SECONDARY OUTCOMES:
Cognitive health status: presence or absence of diagnosed Alzheimer's disease. | Day 1 Just After inclusion
  Spatial navigation strategies will be compared according to participant's cognitive status (cognitively healthy versus Alzheimer's disease).
P-tau217 plasmatic protein assay in pg/mL interpreted in relation to creatinine levels and body mass index. | Day 1 Just After inclusion
  Spatial navigation strategies will be compared according to the p-tau217 plasmatic protein assay. A Simoa (Single Molecule Array for Protein Detection) platform will use commercial kits to carry out the p-tau217 protein assay (Quanterix).
Genotyping of the apolipoprotein E gene: ApoE4 carrier or ApoE4 non carrier. | Day 1 Just After inclusion
  Spatial navigation strategies will be compared according to the genotyping. A molecular biology platform will carry out genotyping for apolipoprotein E

CONTACTS AND LOCATIONS:
Overall Officials: Antoine GARNIER-CRUSSARD, Principal Investigator — HCL
Locations (3):
- France (3):
  - Hôpital des Charpennes, Institut du Vieillissement, Hospices Civils de Lyon, Villeurbanne, Lyon
  - Service de neuro-cognition et neuro-ophtalmologie Hôpital Pierre Wertheimer, Bron
  - Service de médecine du vieillissement - Hôpital Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No